CLINICAL TRIAL: NCT06748248
Title: Effects of Suspension Therapy on Mobility and Balance in Children With Down Syndrome
Brief Title: Suspension Therapy Effects on Mobility and Balance in Down Syndrome
Acronym: STOMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/Sidra Rukhsar
Record Dates: First submitted 2024-11-03; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Down Syndrome (DS)
Keywords: Down syndrome; Suspension Therapy; Universal Exercise Unit; Pediatric Balance Scale; four Square Step Test; 1min Walk Test; Timed up and go test
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: It will be randomized control trial in which non probability convenient sampling will be used. two groups of 3-6 age will be formed in which participants will be randomly divided. Group A will be receive Suspension Therapy. Group B will be receive routine therapy.
Who Masked: Participant
Masking Description: participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suspension therapy (Experimental): Universal Exercise Unit also named Spider cage and Monkey cage. This device will used in this study. This system helps the children to weight shift, more independent movement and assisted movement such as sit to stand, squats and jumping.
  Interventions: Other: suspension Therapy
- Routine Treatment (Other): These routine exercises will consist of stretching exercises (particularly upper and lower body stretches and full body stretches). Stretches will be gentle and avoid bouncing. Hold for each stretch will be 15-30 seconds. Balance and coordination exercises (Walking on balance beams, obstacle courses) will be performed as RPT. The exercise program will gradually increase in intensity in accordance with each participant's functional improvement. These exercises will be carried out 5 days in a week for one hour daily.
  Interventions: Other: Routine Treatment

INTERVENTIONS:
Other: suspension Therapy — suspension therapy for individuals with Down syndrome is an approach that focuses on improving mobility and balance through different activities that will be conducted through universal exercise unit. This method involves organizing individuals with Down syndrome into two groups. Group A will perform Suspension Therapy in addition to routine physical therapy. These routine exercises will consist of stretching exercises (arm raises, chest stretch, leg swings, hamstring stretch, cat-cow poses, starfish stretch), strength and endurance training (like stepping, carrying light weights) and balance training (playing hopscotch and kicking a ball). The exercise program will gradually increase in intensity in accordance with each participant's functional improvement. Suspension Therapy will consist of passive and active postural auto-correction exercises done repeatedly and based on kinesthetic and sensorimotor principles. Repeated corrective movements will be performed.
  Other Names: universal exercise unit
  Arms: suspension therapy
Other: Routine Treatment — Group B will perform routine physical therapy (RPT) alone. These routine exercises will consist of stretching exercises (particularly upper and lower body stretches and full body stretches). Stretches will be gentle and avoid bouncing. Hold for each stretch will be 15-30 seconds. Balance and coordination exercises (Walking on balance beams, obstacle courses) will be performed as RPT. The exercise program will gradually increase in intensity in accordance with each participant's functional improvement. These exercises will be carried out 5 days in a week for one hour daily.
  Data will be assessed by assessor at baseline and at the end of 5th session of treatment (Pre and post).
  Other Names: routine physical Therapy
  Arms: Routine Treatment

SUMMARY:
Down syndrome (DS) is one of the most common congenital disorders. Individuals with Down syndrome present with several impairments such as hypotonia, ligament laxity, decreased muscle strength, insufficient muscular co-contraction, inadequate postural control, and disturbed proprioception. These factors are responsible for the developmental challenges faced by children with Down syndrome. These individuals also present with balance dysfunctions. Neuromuscular and musculoskeletal impairments due to the chromosomal abnormality lead to developmental delay. These children also exhibit poor balance with greater instability and inefficient compensatory mechanisms including altered center of pressure displacement and trunk stiffening that predisposes them to falls. The aim of this study is to determine the Effects of Suspension Therapy (ST) on mobility and balance of children with Down syndrome. Suspension Therapy using Universal exercise Unit (UEU) is a three dimensional (3D) cage, consists of system of pulleys, suspensions, belts for supporting and elastic cords. Suspension Therapy is based on the concept of unloading the body against gravity and to perform movement of weak part of body.

DETAILED DESCRIPTION:
The current study will be Randomized Controlled Trial. Inclusion criteria for the study will be children with Down syndrome (DS) of mild to moderate mental retardation aged between 3 and 6 years. Patients with any cardiac issue and orthopedic limitation to exercise such as hip, knee, foot or spinal deformities will be excluded from the study. A sample of 26 children with DS will be selected from both genders. Tools used for data collection will be Pediatric Balance scale (PBS), Four square step test (FSST), Timed up and Go test (TUG) and 1Minute Walk Test (1MWT). Participants will be measured before and after treatment to assess changes. Interventions are carried out 5 days in a week for one hour daily. In this study descriptive statistical tools will used to analyze the data. Data will be analyzed through SPSS version 23.00.

ELIGIBILITY:
Inclusion Criteria: • Diagnosed children with Down syndrome with mild (IQ: 69-50) to moderate (IQ: 50-35) mental retardation

* Aged between 3 to 6 years
* Both gender
* Able to follow the instructions
* Able to stand and walk

Exclusion Criteria: • Any Cardiovascular disease

* Visual and Hearing impairment
* Orthopedic limitation to exercise such as hip, knee, foot or spinal deformities

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
1 Minute Walk Test | 1 minute
  The distance covered during the 1 minute walk test was compared with the children gross motor function as assessed by the Gross Motor Function Measure. We concluded that the 1 Minute Walk Test is a valid measure for assessing functional ability in children with bilateral spastic cerebral palsy. Its cost effectiveness and user friendliness make it a potentially useful tool in the clinical setting. The test retest reliability of a 1 minute walk test at a child maximum walking speed was assessed in children with bilateral spastic cerebral palsy. A 1 minute walk test is a reliable method of assessing function in children with Cerebral palsy but care must be taken when interpreting changes in individual patient data.
Four Square Step Test | 15 seconds
  Four Square Step Test is a tool for measuring balance in children with Down syndrome by stepping over four squares. The Four Square Step Test is a balance and mobility assessment that evaluates a persons ability to step quickly and accurately in multiple directions. Participants step in and out of four squares arranged in a cross pattern starting from one of the outer squares and moving through a sequence. The test is timed and results help identify balance impairments and fall risks. A completion time of under 15 seconds is generally considered normal.

SECONDARY OUTCOMES:
Pediatric balance scale | 15 to 20 minutes
  The Pediatric Balance Scale a modification of the Berg Balance Scale will be used as a balance measure for children. The pediatric balance scale measure can be performed without specialized equipment and is quickly and easily administered. The Pediatric balance scale has been used to measure the balance functions for school age children with mild to moderate motor impairment and children with Cerebral palsy. The tasks range from timed sitting balance to standing on one leg. This study confirmed good validity of the Pediatric balance scale and its capability to predict motor function and Activity of daily living at follow up. The Pediatric balance scale static dynamic and total were moderately responsive to change.
Timed Up and Go Test | The Timed Up and Go Test typically takes about 5 to 10 minutes to complete. This includes time for instructions the actual test which usually lasts 10 to 30 seconds depending on the individual and scoring.
  The Timed Up and Go Test is a quick assessment used to evaluate mobility and balance primarily in older adults. It measures the time it takes for a participant to stand up from a chair walk 3 meters or 10 feet turn around walk back and sit down. The total time is recorded with results helping to identify fall risk and assess functional mobility. A completion time under 10 seconds is typically considered normal while over 12 seconds may indicate an increased risk of falls.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Rukhsar, MS, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Riphah International University, Lahore, Punjab Province
  - Riphah International Universiy, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendez-Martinez M, Rodriguez-Grande EI. Effects of therapeutic exercise on the motor function of adults with Down syndrome: a systematic review and meta-analysis. Sci Rep. 2023 Dec 11;13(1):21962. doi: 10.1038/s41598-023-48179-1. PMID 38081839